CLINICAL TRIAL: NCT03944096
Title: Efficacy and Safety of Faecal Microbiota Transplantation in Patients With Rheumatoid Arthritis Refractory to Methotrexate: a 24-week, Double-Blind, Randomised Trial
Brief Title: Efficacy and Safety of Fecal Microbiota Transplantation in Patients With Rheumatoid Arthritis Refractory to Methotrexate
Acronym: FARM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Xuan Zhang, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FARM
Record Dates: First submitted 2019-05-08; First posted 2019-05-09 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Rheumatoid Arthritis
Keywords: fecal microbiota transplantation; methotrexate; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT+MTX (Experimental): FMT One FMT is performed at baseline by gastroscopic guidance. The same FMT is repeated 4 weeks later. The transplant consists of 50 g mixed feces obtained from 3-5 non-related healthy donors. The donor feces is suspended into NaCl (0.9%) and glycerol (10%), and will be stored at minus 80 degrees celsius until use. The total volume of the suspension is 150 mL and its temperature will be 37 degrees celsius when infused into ileus of the recipient.
  Drug: Methotrexate (MTX) Weekly methotrexate
  Interventions: Procedure: FMT+MTX
- autologous FMT+MTX (Placebo Comparator): autologous FMT (the feces used in FMT is from participant themselves) One identical FMT is performed at baseline using gastroscopic guidance and is repeated 4 weeks later. The corresponding participant's feces is suspended into NaCl (0.9%) and glycerol (10%), and will be stored at minus 80 degrees celsius until use. The total volume of the suspension is 150 mL and its temperature will be 37 degrees celsius when infused into ileus of the participant himself or herself.
  Drug: Methotrexate (MTX) Weekly methotrexate
  Interventions: Procedure: FMT+MTX

INTERVENTIONS:
Procedure: FMT+MTX — FMT is performed at the beginning of the study and is repeated after 4 weeks plus MTX in the same dose.

SUMMARY:
In this 24-week, single center, randomized, double-blind study, the investigators will evaluate the efficacy and safety of fecal microbiota transplantation in patients with active rheumatoid arthritis refractory to methotrexate

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic autoimmune disease, characterized by painful synovium inflammation, bony erosions, immune activation. Gut microbiota plays an important role in pathophysiology of RA. FMT(fecal microbiota transplantation) is the engraftment of microbiota from a healthy donor into a recipient to achieve restoration of the normal gut microbial community structure.This study evaluates the efficacy and safety of FMT with methotrexate in patients with active RA refractory to methotrexate

Objectives:

1. To evaluate the efficacy of FMT with MTX for the treatment of signs and symptoms of RA in patients refractory to MTX.
2. To evaluate the safety of FMT with MTX for the treatment of signs and symptoms of RA in patients refractory to MTX DESIGN

This is a Phase 2, randomized, 24-week, double-blind, parallel group study, and 30 patients with active RA refractory to MTX will be randomized in a 1:1 ratio to one of the following 2 parallel treatment arms:

1. FMT from healthy donor plus methotrexate
2. autologous FMT(from the participant himself/herself) plus methotrexate

Escape:

On week 16, all participants with inadequate response, defined as a <20% improvement of swollen and tender joint counts from baseline can switch type and dose of DMARDs.

Endpoints :

1. Primary endpoint:

   ACR20 response rates at 16 weeks.
2. Secondary endpoint： 1）ACR50 and ACR70 response at 16, 24 weeks，ACR20 response at 24 weeks. 2）DAS 28 (CRP) and DAS 28 (ESR) at 16 and 24 weeks. 3) EULAR response rates at 16 and 24 weeks. 4) Health assessment questionnaire (HAQ) at 16 and 24 weeks. 5) Patient assessment of arthritis pain at 16 and 24 weeks. 6) Patient and physician global assessment of arthritis at 16 and 24 weeks

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years with informed consent
* Fulfill the 2010 ACR/EULAR classification criteria for rheumatoid arthritis
* Positive RF or anti-CCP antibody on screening
* Have active RA shown by swollen joint count(SJC)≥4 and tender joint count(TJC)≥4 and ESR >28 mm/hr or C-reactive protein > 1.5 ULN
* Have received methotrexate for 3 months or longer and at a stable dose of 7.5 to 25 mg/week (extremes included) for at least four weeks prior to screening and willing to continue on this regimen for the duration of the study.
* Class I, II or III of the ACR 1991 Revised Criteria for Global Functional Status in RA
* If taking oral steroids, these should be at a dose ≤10 mg/day of prednisone or prednisone equivalent and stable for at least four weeks prior to screening;
* If taking non-steroidal anti-inflammatory drugs (NSAIDs), these must be at a stable dose for at least two weeks prior to screening;
* Female subjects must have a negative pregnancy test unless they are surgically sterile or have been post-menopausal for at least one year (12 consecutive months without menses);
* Women of childbearing potential must use a medically acceptable means of birth control and agree to continue its use during the study and for at least four weeks after the last dose of study drug. Sexually active men must agree to use a medically acceptable form of contraception during the study and continue its use for at least 3 months after the last dose of study drug; and
* Willing to suspend the use of other adjuvant treatment for the duration of the study including acupuncture, massage, etc.

Exclusion Criteria:

* Pregnant, lactating or further fertility requirements
* History of any inflammatory rheumatological disorders other than RA;
* Previously received any biologic agents.
* Treatment with disease-modifying antirheumatic drugs (DMARDs), other than background methotrexate;
* Receipt of an intra-articular or parenteral corticosteroid injection within four weeks prior to screening;
* Active or chronic infection, including HIV, HCV, HBV, tuberculosis.
* Malignancy or history of malignancy.
* Severe, progressive, or uncontrolled cardiac, pulmonary, renal, hepatic, gastrointestinal, hematologic, metabolic, endocrine or neurologic disease
* unable to undergo colonoscopy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
The American College of Rheumatology 20 (ACR20) response at 16 weeks | week 16
  The difference of ACR20 between Arm 1 (FMT+MTX) and Arm 2 (autologous FMT+MTX)

SECONDARY OUTCOMES:
The American College of Rheumatology 50/70 (ACR50/ACR70) response at 16 weeks | week 16
  The difference of ACR50/70 between Arm 1 (FMT+MTX) and Arm 2 (autologous FMT+MTX)
The American College of Rheumatology 20/50/70 (ACR20/ACR50/ACR70) response at 24 weeks | week 24
  The difference of ACR20, ACR50 and ACR70 between Arm 1 (FMT+MTX) and Arm 2(autologous FMT+MTX) at week 24
The Disease Activity Score-28 (DAS28) response at 16 weeks | week 16
  The change in DAS28 score from baseline to week 16 between Arm 1 (FMT+MTX) and Arm 2(autologous FMT+MTX).
  DAS28 ＝ 0.56*SQRT(TJC28) + 0.28*SQRT(SJC28) + 0.36*ln(CRP + 1) + 0.014*GH + 0.96 TJC28: The number of tender joints (0-28). SJC28: The number of swollen joints (0-28). CRP: The C-Reactive Protein level (in mg/l). GH: The patient global health assessment (from 0=best to 100=worst). The 28 joint: shoulders, elbows, wrists, metacarpophalangeal joints, proximal interphalangeal joints and the knees.
The Disease Activity Score-28 (DAS28) response at 24 weeks | week 24
  The change in DAS28 score from baseline to week 24 between Arm 1 (FMT+MTX) and Arm 2(autologous FMT+MTX).
  DAS28 ＝ 0.56*SQRT(TJC28) + 0.28*SQRT(SJC28) + 0.36*ln(CRP + 1) + 0.014*GH + 0.96 TJC28: The number of tender joints (0-28). SJC28: The number of swollen joints (0-28). CRP: The C-Reactive Protein level (in mg/l). GH: The patient global health assessment (from 0=best to 100=worst). The 28 joint: shoulders, elbows, wrists, metacarpophalangeal joints, proximal interphalangeal joints and the knees.
The European League Against Rheumatism (EULAR) response at 16 weeks | week 16
  The difference of proportions of patients meeting EULAR response between Arm 1(FMT+MTX) and Arm 2 (autologous FMT+MTX) at week 16
Health Assessment Questionnaire without Didability Index (HAQ-DI) at 16 weeks | week 16
  The change in HAQ-DI score from baseline to week 16 between Arm 1(FMT+MTX) and Arm 2 (autologous FMT+MTX).
  HAQ-DI is an index measuring the quality of life related to health, which includes 20 questions in terms of three categories:
  from 0 to 1: mild difficulties to moderate disability, from 1 to 2: disability moderate to severe, from 2 to 3: severe to very severe disability. The mean score is recorded as the result.
Incidence of adverse events and sever adverse events (SAE) during the study | week 24
  Safety profile

CONTACTS AND LOCATIONS:
Overall Officials: Xuan Zhang, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided